CLINICAL TRIAL: NCT00123279
Title: A Dose-escalation Clinical Trial of Intravitreal Microplasmin in Patients Undergoing Surgical Vitrectomy for Vitreomacular Traction Maculopathy
Brief Title: Intravitreal Microplasmin in Patients Undergoing Surgical Vitrectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Responsible Party: Edith Van Dijkman, ThromboGenics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG-MV-001
Record Dates: First submitted 2005-07-21; First posted 2005-07-22 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Vitreomacular Traction Maculopathy; Eye Diseases
Keywords: diabetic macular edema; macular hole; vitreomacular traction syndrome
MeSH Terms: conditions — Eye Diseases; Retinal Perforations | interventions — microplasmin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Experimental)
  Interventions: Drug: Microplasmin
- 2 (Experimental)
  Interventions: Drug: Microplasmin
- 3 (Experimental)
  Interventions: Drug: Microplasmin
- 4 (Experimental)
  Interventions: Drug: Microplasmin
- 5 (Experimental)
  Interventions: Drug: Microplasmin
- 6 (Experimental)
  Interventions: Drug: Microplasmin

INTERVENTIONS:
Drug: Microplasmin — 25ug injected 1 hr prior to PPV, 24 hr and 7 days prior to PPV, 50ug injected 24 hr prior to PPV, 75ug injected 24 hr prior to PPV and 125ug injected 24 hr prior to PPV.

SUMMARY:
The purpose of this trial is to evaluate the safety and preliminary efficacy of different doses and several exposure times of intravitreal microplasmin in the setting of pars plana vitrectomy for vitreomacular traction maculopathy.

DETAILED DESCRIPTION:
Study drug will be administered in the mid-vitreous by injection. Patients will be enrolled into the cohorts in a sequential dose/time-escalating fashion. To ensure that enrolment is evenly balanced across eligible conditions, enrolment of any specific underlying disease type into any cohort will be capped at five (5) patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with vitreomacular traction maculopathy for whom vitrectomy is indicated, according to the principal investigator, including:

  * Macular edema associated with vitreomacular traction (DME, VMTS);
  * Stage II-III macular hole of < 6 months duration since symptom onset;
  * Demonstration of vitreomacular adhesion (based on preoperative optic coherence tomography [OCT]) in the study eye;
  * OCT - presence of posterior hyaloid membrane inserting on to the macula, but with some area of clear separation visible between the retina and the posterior hyaloid.

Exclusion Criteria:

* Evidence of fibrocellular proliferation characterized by whitish epimacular tissue (surface wrinkling is not an exclusion criterion).
* Patients with vitreous hemorrhage which precludes either of the following: visualization of the posterior pole by visual inspection OR adequate assessment of the macula by either OCT and/or fluorescein angiogram in the study eye.
* Patients with rhegmatogenous retinal detachment, proliferative vitreoretinopathy (PVR), or retinal degenerative changes in the study eye.
* Patients with high myopia or aphakia in the study eye
* Patients with history of rhegmatogenous retinal detachment in the fellow eye or family history of retinal detachment
* Patients who are considered likely to require intraocular surgery in the study eye for any reason other than vitreomacular traction maculopathy/macular edema in the coming three months.
* Patients who have had ocular surgery in the study eye in the prior three months.
* Patients who have had a vitrectomy in the study eye at any time.
* Patients with a history of uveitis or significant trauma in the study eye.
* Patients who are currently being treated for glaucoma in the study eye.
* Patients who have had laser photocoagulation treatment in the study eye in the previous 3 months.
* Intravitreal injection of any drug in the study eye in the previous 6 months or during the study.
* Patients who are pregnant or of child-bearing potential not utilizing a form of contraception acceptable to the investigator.
* Patients who, in the investigator's view, will not complete all visits and investigations, including the exit visit at 6 months.
* Patients who have participated in an investigational drug study within the past 30 days.
* HgA1c > 9%.
* Patients with hypertension (either systolic blood pressure [SBP] > 170 or diastolic blood pressure [DBP] > 100 mm Hg).
* Patients with a life-expectancy less than 6 months.
* Patients who have previously participated in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-12; Primary Completion 2007-02 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Grade of Posterior Vitreous Detachment (PVD) preoperatively and release of vitreomacular traction | Baseline, 1,2 and 3hr, 1, 3, 14, 28, 90 and 180 Days

SECONDARY OUTCOMES:
The occurrence of any (serious) adverse event | Throught-out the study

CONTACTS AND LOCATIONS:
Overall Officials: Marc deSmet, Prof. Dr, Principal Investigator — Amsterdam UMC, location VUmc
Locations (3):
- University Hospital Gasthuisberg, Leuven, Belgium
- Netherlands (2):
  - Academic Medical Center, University of Amsterdam, Amsterdam
  - Oogziekenhuis Rotterdam, Rotterdam